CLINICAL TRIAL: NCT02489942
Title: Post Marketing Surveillance in Japan on Long Term Drug Use of JARDIANCE® Tablets in Patients With Type 2 Diabetes Mellitus
Brief Title: Long Term Daily Use of JARDIANCE® Tablets in Japanese Patients With Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245.94
Record Dates: First submitted 2015-05-21; First posted 2015-07-03 (Estimated); Results first posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2021-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Jardiance: Patients with T2DM to receive Jardiance tablets 10 mg, 25 mg
  Interventions: Drug: Jardiance

INTERVENTIONS:
Drug: Jardiance — Empagliflozin

SUMMARY:
Study to investigate the safety and efficacy of long-term daily use of JARDIANCE® Tablets in Japanese patients with type 2 diabetes mellitus

ELIGIBILITY:
Inclusion criteria:

Male and female Japanese patients with type 2 diabetes mellitus who have never been treated with JARDIANCE® Tablets before the enrolment

Exclusion criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3,000 Japanese patients with the assessment of 3-year completed administration
Sampling Method: Non-Probability Sample
Enrollment: 8145 (Actual)
Dates: Start 2015-06-12 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Multiple Locations, Japan

REFERENCES:
- [Derived] Kaku K, Chin R, Naito Y, Iliev H, Ikeda R, Ochiai K, Yasui A. Safety and effectiveness of empagliflozin in Japanese patients with type 2 diabetes: interim analysis from a post-marketing surveillance study. Expert Opin Drug Saf. 2020 Feb;19(2):211-221. doi: 10.1080/14740338.2020.1694659. Epub 2019 Nov 26. PMID 31769309
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A non-interventional study to investigate the safety and efficacy of longterm daily use of JARDIANCE® Tablets in Japanese patients with type 2 diabetes mellitus.
Pre-assignment Details: Non-randomized, post marketing surveillance, a prospective study using a continuous investigation system. No specific criteria (e.g. demographic, baseline concomitant drug in use) were defined for participant enrollment.
Groups:
- JARDIANCE® User 10 Milligram (mg) or 25 mg: Japanese patients with type 2 diabetes mellitus (T2DM) who never received JARDIANCE® before enrollment and who completed a 3-year JARDIANCE® observation period between June 2015 and November 2020. The usual dose was 10 milligrams (mg) of a JARDIANCE® tablet administered orally once daily. If the treatment effectiveness was insufficient, the daily dose could be increased to 25 mg once daily while the patient's condition was being carefully monitored. Duration of treatment was up to 246 weeks.
Period: Overall Study
Arm/Group | JARDIANCE® User 10 Milligram (mg) or 25 mg
Started | 8145
Case Report Form (CRF) Collected | 8059
Treated | 8057
Completed | 4729
Not Completed | 3416
Not completed — Request by patient | 602
Not completed — Improvement/remission | 157
Not completed — No change/Progressive disease | 263
Not completed — Adverse Event | 522
Not completed — Other personal reasons | 1218
Not completed — Lost to Follow-up | 456
Not completed — Not continuously investigated | 7
Not completed — Patient started jardiance treatment out of registration period | 1
Not completed — Multiple registration | 1
Not completed — No patient visit after entry | 100
Not completed — No treatment with Jardiance | 2
Not completed — Patient received Jardiance before registration | 1
Not completed — No CRF collected | 86

BASELINE CHARACTERISTICS:
Population: Safety Set: All patients who had received treatment of JARDIANCE® tablet at least one time except those who were found to have no observation after enrollment, invalid registration, or invalid contract with the site.
Arm/Group | JARDIANCE® User 10 Milligram (mg) or 25 mg
Number analyzed (Participants) | 7947
Age, Continuous [Mean (Standard Deviation); unit: Years] — Safety Set.
  Years | 58.8 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Set
  Participants
    Female | 2939
    Male | 5008
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Drug Reactions (ADRs)
Description: Number of patients with adverse drug reactions.
Time Frame: From first drug administration until 7 days after last drug administration, up to 247 weeks.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | JARDIANCE® User 10 Milligram (mg) or 25 mg
Number analyzed (Participants) | 7947
Participants | 1029

2. Secondary Outcome: Change From Baseline in Haemoglobin A1c (HbA1c) at the Last Observation During the Observation Period
Description: Change from baseline in haemoglobin A1c (HbA1c) at the last observation during the observation period.
Time Frame: At start of treatment and at last observation on treatment, up to 246 weeks.
Population: Efficacy set: All patients in the safety set, except patients who had no available efficacy data and/or do not suffer from type 2 diabetes mellitus.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | JARDIANCE® User 10 Milligram (mg) or 25 mg
Number analyzed (Participants) | 7314
Percentage change | -0.74 (1.34)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at the Last- Observation During Observation Period
Description: Change from baseline in fasting plasma glucose (FPG) at the last- observation during observation period.
Time Frame: At start of treatment and at last observation on treatment, up to 246 weeks.
Population: All patients included in the efficacy set and with available data for this endpoint.
Measure: Mean (Standard Deviation); unit: Milligram/deciliter (mg/dL)
Arm/Group | JARDIANCE® User 10 Milligram (mg) or 25 mg
Number analyzed (Participants) | 2510
Milligram/deciliter (mg/dL) | -30.1 (55.5)

ADVERSE EVENTS:
Time Frame: From first drug administration until 7 days after last drug administration, up to 247 weeks.
Description: Safety Set: All patients who had received treatment of JARDIANCE Tablet at least one time except those who were found to have no observation after enrolment, invalid registration, or invalid contract with the site.
Arm/Group | JARDIANCE® User 10 Milligram (mg) or 25 mg
All-Cause Mortality (participants affected / at risk) | 42/7947
Serious Adverse Events (participants affected / at risk) | 381/7947
Other Adverse Events (participants affected / at risk) | 0/7947
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JARDIANCE® User 10 Milligram (mg) or 25 mg (N=7947)
Anaemia (Blood and lymphatic system disorders) | 3
Pancytopenia (Blood and lymphatic system disorders) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 19
Acute myocardial infarction (Cardiac disorders) | 13
Cardiac failure (Cardiac disorders) | 9
Myocardial infarction (Cardiac disorders) | 7
Atrial fibrillation (Cardiac disorders) | 3
Cardiac failure congestive (Cardiac disorders) | 3
Sinus node dysfunction (Cardiac disorders) | 3
Coronary artery stenosis (Cardiac disorders) | 2
Ventricular extrasystoles (Cardiac disorders) | 2
Adams-Stokes syndrome (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Bundle branch block bilateral (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Prinzmetal angina (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Intracardiac thrombus (Cardiac disorders) | 1
Silent myocardial infarction (Cardiac disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Congestive cardiomyopathy (Cardiac disorders) | 1
Phimosis (Congenital, familial and genetic disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 3
Deafness neurosensory (Ear and labyrinth disorders) | 2
Deafness (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Glaucoma (Eye disorders) | 3
Diabetic retinopathy (Eye disorders) | 2
Cataract (Eye disorders) | 1
Cataract diabetic (Eye disorders) | 1
Eyelid ptosis (Eye disorders) | 1
Posterior capsule opacification (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Macular hole (Eye disorders) | 1
Normal tension glaucoma (Eye disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 3
Melaena (Gastrointestinal disorders) | 2
Autoimmune pancreatitis (Gastrointestinal disorders) | 2
Acute abdomen (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Salivary gland calculus (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Sudden death (General disorders) | 4
Chest pain (General disorders) | 2
Chest discomfort (General disorders) | 1
Death (General disorders) | 1
Fatigue (General disorders) | 1
Inflammation (General disorders) | 1
Vascular stent stenosis (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Cholangitis (Hepatobiliary disorders) | 3
Cholelithiasis (Hepatobiliary disorders) | 3
Bile duct stone (Hepatobiliary disorders) | 2
Cholangitis acute (Hepatobiliary disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 2
Biliary colic (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hepatitis alcoholic (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Bile duct stenosis (Hepatobiliary disorders) | 1
Liver injury (Hepatobiliary disorders) | 1
Biliary obstruction (Hepatobiliary disorders) | 1
Immune system disorders (Hepatobiliary disorders) | 1
Anaphylactic shock (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 10
Pneumonia (Infections and infestations) | 4
Pyelonephritis (Infections and infestations) | 4
Diabetic gangrene (Infections and infestations) | 3
Appendicitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Infection (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Pneumonia bacterial (Infections and infestations) | 2
Brain abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Endometritis (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Genital herpes (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Osteomyelitis chronic (Infections and infestations) | 1
Pneumonia mycoplasmal (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Lymph gland infection (Infections and infestations) | 1
Beta haemolytic streptococcal infection (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Acute hepatitis B (Infections and infestations) | 1
Abdominal abscess (Infections and infestations) | 1
Tonsillitis bacterial (Infections and infestations) | 1
Emphysematous pyelonephritis (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1
Complicated appendicitis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 13
Road traffic accident (Injury, poisoning and procedural complications) | 6
Subdural haematoma (Injury, poisoning and procedural complications) | 4
Fibula fracture (Injury, poisoning and procedural complications) | 3
Humerus fracture (Injury, poisoning and procedural complications) | 3
Tibia fracture (Injury, poisoning and procedural complications) | 3
Upper limb fracture (Injury, poisoning and procedural complications) | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 2
Fracture (Injury, poisoning and procedural complications) | 2
Joint dislocation (Injury, poisoning and procedural complications) | 2
Rib fracture (Injury, poisoning and procedural complications) | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 2
Heat illness (Injury, poisoning and procedural complications) | 2
Adrenal gland injury (Injury, poisoning and procedural complications) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Suture rupture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Brain contusion (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1
Blood glucose increased (Investigations) | 2
Blood pressure decreased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Glycosylated haemoglobin increased (Investigations) | 1
Weight increased (Investigations) | 1
Brain natriuretic peptide increased (Investigations) | 1
Metabolism and nutrition disorders (Investigations) | 30
Diabetes mellitus inadequate control (Investigations) | 12
Hyperglycaemia (Investigations) | 5
Diabetes mellitus (Investigations) | 4
Hypoglycaemia (Investigations) | 3
Dehydration (Investigations) | 2
Diabetic ketosis (Investigations) | 1
Ketoacidosis (Investigations) | 1
Marasmus (Investigations) | 1
Dyslipidaemia (Investigations) | 1
Decreased appetite (Investigations) | 1
Musculoskeletal and connective tissue disorders (Investigations) | 12
Osteoarthritis (Investigations) | 5
Arthralgia (Investigations) | 1
Fracture malunion (Investigations) | 1
Lumbar spinal stenosis (Investigations) | 1
Muscle spasms (Investigations) | 1
Polymyalgia rheumatica (Investigations) | 1
Rhabdomyolysis (Investigations) | 1
Rotator cuff syndrome (Investigations) | 1
Spinal stenosis (Investigations) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 20
Dementia (Nervous system disorders) | 5
Epilepsy (Nervous system disorders) | 3
Carotid artery stenosis (Nervous system disorders) | 2
Cerebellar infarction (Nervous system disorders) | 2
Cerebral haemorrhage (Nervous system disorders) | 2
Myelopathy (Nervous system disorders) | 2
Subarachnoid haemorrhage (Nervous system disorders) | 2
Lacunar infarction (Nervous system disorders) | 2
Thalamus haemorrhage (Nervous system disorders) | 2
Thrombotic cerebral infarction (Nervous system disorders) | 2
Altered state of consciousness (Nervous system disorders) | 1
Brain stem haemorrhage (Nervous system disorders) | 1
Brain stem infarction (Nervous system disorders) | 1
Cerebellar atrophy (Nervous system disorders) | 1
Cerebral atrophy (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Moyamoya disease (Nervous system disorders) | 1
Multiple sclerosis (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Neuralgic amyotrophy (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Cerebral haematoma (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Embolic cerebral infarction (Nervous system disorders) | 1
Parkinson's disease (Nervous system disorders) | 1
Generalised onset non-motor seizure (Nervous system disorders) | 1
Schizophrenia (Psychiatric disorders) | 2
Completed suicide (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Psychiatric symptom (Psychiatric disorders) | 1
Cardiovascular somatic symptom disorder (Psychiatric disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 2
Calculus urinary (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal artery stenosis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Pyelocaliectasis (Renal and urinary disorders) | 1
Ureterolithiasis (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Cystocele (Reproductive system and breast disorders) | 1
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1
Ovarian haemorrhage (Reproductive system and breast disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1
Knee operation (Surgical and medical procedures) | 1
Enterostomy (Surgical and medical procedures) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2
Aneurysm (Vascular disorders) | 1
Aortic dissection (Vascular disorders) | 1
Varicose vein (Vascular disorders) | 1
Lymphocele (Vascular disorders) | 1
Hypertensive emergency (Vascular disorders) | 1
Infarction (Vascular disorders) | 1
Arterial occlusive disease (Vascular disorders) | 1
Peripheral venous disease (Vascular disorders) | 1
Subclavian vein occlusion (Vascular disorders) | 1
Device occlusion (Product Issues) | 1

LIMITATIONS AND CAVEATS:
Since this surveillance was an observational, non interventional study, it lacked the methodological rigour of a randomised control trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-04-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT02489942/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT02489942/SAP_001.pdf